CLINICAL TRIAL: NCT04010838
Title: Effectiveness Research for Severe Disorders of Consciousness Patients Treated With Spinal Cord Stimulation (SCS)
Brief Title: Spinal Cord Stimulation in Patients With Disorders of Consciousness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xuehai Wu, Professor, Huashan Hospital, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2017-329
Record Dates: First submitted 2019-05-18; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Disorder of Consciousness; Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; spinal cord stimulation; DoC; SCS
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Random controlled trial
Who Masked: Outcomes Assessor
Masking Description: People who involved with data analysis and outcomes assessment would be blind to the randomization procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (No Intervention)
- Spinal cord stimulation and conventional treatment (Experimental)
  Interventions: Procedure: spinal cord stimulation

INTERVENTIONS:
Procedure: spinal cord stimulation — The spinal cord stimulation(SCS) is a type of implantable neuromodulation device (spinal cord stimulator) that is used to send electrical signals to select areas of the spinal cord (C2-C4 in this study) for the treatment of disorders of consciousness.
  Arms: Spinal cord stimulation and conventional treatment

SUMMARY:
Disorders of consciousness(DOC) is the most serious complications and has been widely paid attention to by the government. DOC patients cause large social and economic burden to our society for there has no effective cure so far. Spinal cord stimulation(SCS) for wake-promoting therapy has aroused scholars' attention and become a hot area recently. There was much debate about the effectiveness of SCS therapy, but because of the limitation of our understanding of consciousness and the uncertainty of parameters of the stimulation, So, to figure out the indications and effectiveness of neuromodulation therapy should be the first step, and finding individual treatment and parameter may have important implications for DOC patients.

DETAILED DESCRIPTION:
The spinal cord stimulation therapy is explorative at best at the moment. Attempts to improve the level of consciousness of patients in the different stages of DOC have shown some promise. Spinal cord stimulation(SCS) seem promising in some studies, suggesting that further research is needed. Current publications of DOC spinal cord stimulation therapy was not convincing because of the small number of patients and no randomized controlled trial. Therefore, there was much debate about the effectiveness of spinal cord stimulation therapy because of the limitation of our understanding of consciousness and the uncertainty of parameters of neuromodulation. The better understanding of brain function and large randomized trials are necessary. Future research should also focus on identifying specific neuro-biomarkers (i.e. neural network). So, to figure out the indications and effectiveness of neuromodulation therapy should be the first step, and finding individual treatment and parameter may have important implications for DOC patients.

Scientific Issues Targeted:1) To figure out the effectiveness of spinal cord stimulation therapy using random controlled trial. 2) To explore individual parameters of SCS techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14 to 65 years old;
2. DOC patients, including vegetative state and minimally consciousness state.
3. With normal body temperature, stable vital signs, spontaneous breathing without an extra oxygen supply, no tracheotomy using metal trachea cannula, and feasible for magnetic resonance inspectors;
4. Written informed consent from patient families

Exclusion Criteria:

1. History of nervous or spirit disorders, or some other serious diseases such as cardiac or pulmonary problems;
2. With contraindications of spinal cord operations.
3. Body temperature is abnormal, vital signs are not stable, still need a ventilator to support breathing; Plentiful sputum needed suction during MRI scans.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
the JFK Coma Recovery Scale-Revised (CRS-R) scale | at baseline (T0), which means 1 month before stimulation.
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.
the JFK Coma Recovery Scale-Revised (CRS-R) scale | 2 weeks after the end of the treatment (T1)
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.
the JFK Coma Recovery Scale-Revised (CRS-R) scale | 3 months after the end of the treatment (T2)
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.
the JFK Coma Recovery Scale-Revised (CRS-R) scale | 6 months after the end of the treatment(T3)
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.

SECONDARY OUTCOMES:
EEG recording in resting state with Phase Coherence analysis(PC index) | at baseline (T0), which means 1 month before stimulation.
  EEG data will be collected using a 256-channel EEG recording system(GES300, Electrical Geodesic, Inc., USA). Phase Coherence index will be performed in MATLAB by first taking the phase of the spectral signals(A), and the caculating as the following: mean[cos(A),2]^2 + mean[sin(A),2]^2
EEG recording in resting state with Phase Coherence analysis(PC index) | 2 weeks after the end of the treatment (T1)
  EEG data will be collected using a 256-channel EEG recording system(GES300, Electrical Geodesic, Inc., USA). Phase Coherence index will be performed in MATLAB by first taking the phase of the spectral signals(A), and the caculating as the following: mean[cos(A),2]^2 + mean[sin(A),2]^2
EEG recording in resting state with Phase Coherence analysis(PC index) | 3 months after the end of the treatment (T2)
  EEG data will be collected using a 256-channel EEG recording system(GES300, Electrical Geodesic, Inc., USA). Phase Coherence index will be performed in MATLAB by first taking the phase of the spectral signals(A), and the caculating as the following: mean[cos(A),2]^2 + mean[sin(A),2]^2
EEG recording in resting state with Phase Coherence analysis(PC index) | 6 months after the end of the treatment (T3)
  EEG data will be collected using a 256-channel EEG recording system(GES300, Electrical Geodesic, Inc., USA). Phase Coherence index will be performed in MATLAB by first taking the phase of the spectral signals(A), and the caculating as the following: mean[cos(A),2]^2 + mean[sin(A),2]^2

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Huashan Hospital, Shanghai, Shanghai Municipality, China